CLINICAL TRIAL: NCT01037231
Title: A Phase 2/3, Double-blind, Randomized, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of OxabactTM to Reduce Urinary Oxalate in Subjects With Primary Hyperoxaluria.
Brief Title: Phase 2/3 Oxabact Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: OxThera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OC3-DB-02
Record Dates: First submitted 2009-12-18; First posted 2009-12-22 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Primary Hyperoxaluria
Keywords: hyperoxaluria; oxalate; PH
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxabact (tm) (Experimental)
  Interventions: Biological: Oxalobacter formigenes
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Oxalobacter formigenes — NLT (not less than) 10^7 CFU oxalobacter formigenes twice daily for 24 weeks
  Other Names: Oxabact; OC3
  Arms: Oxabact (tm)
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Oxalobacter formigenes is effective at lowering urinary oxalate levels in patients with primary hyperoxaluria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (as applicable for the age of the subject)
2. Male or female subjects ≥ 2 years of age
3. A mean urinary oxalate excretion of > 1.0 mmol/1.73m2/day from eligible urine collections performed during screening.
4. A diagnosis of PH I or PH II by one of the following:

   1. Liver biopsy confirmation of deficient liver specific peroxisomal alanine-glyoxylate aminotransferase, (AGT) or mislocalization of AGT from peroxisomes to mitochondria (PH I) or deficient glyoxylate reductase/hydroxypyruvate reductase (GRHPR) activity (PH II)
   2. Homozygosity or compound heterozygosity for a known mutation in the causative genes for PH I and PH II.
   3. Increased glycolate excretion for PH I or increased L-glycerate excretion for PH II.
5. Subjects receiving pyridoxine must be receiving a stable dose for at least 3 months prior to entry into the study and must remain on the stable dose during the study. Subjects not receiving pyridoxine at study entry must be willing to refrain from initiating pyridoxine during study participation.
6. Renal function defined as an estimated GFR ≥ 40 ml/min normalized to 1.73m2 body surface area, or a creatinine clearance of ≥ 40 ml/min normalized to 1.73m2 body surface area.

   Exclusion Criteria:
7. Inability to collect two complete 24-hour urine samples. Each urine collection will be evaluated for completeness based on the urine acceptance criteria outlined in section 11.1.
8. Subjects diagnosed as PH I who are pyridoxine naïve.
9. Subjects that have undergone transplantation (solid organ or bone marrow).
10. The existence of secondary hyperoxaluria, e.g. chronic gastrointestinal diseases such as cystic fibrosis, chronic inflammatory bowel disease and short-bowel syndrome.
11. Current systemic (oral, IM, IV) antibiotic use or received systemic antibiotics within 14 days of study enrolment.
12. History of a recurrent infection requiring >2 courses of systemic antibiotics in the past 6 months, or chronic antimicrobial suppression.
13. Subjects who require immune suppressive therapy (including prednisone > 10mg daily for more than 2 weeks).
14. Current treatment with a separate ascorbic acid preparation. Ascorbic acid up to 250mg/day as a component of a multivitamin formulation is not excluded.
15. Known hypersensitivity to esomeprazol (or any of the other ingredients of this medicine), or to any other proton pump inhibitor medicine. (Nexium contraindication)
16. Concomitant treatment with atazanavir. (Nexium contraindication)
17. Pregnancy.
18. Women of child-bearing potential who are not using adequate contraceptive precautions. Sexually active females, unless surgically sterile or at least 2 years post-menopausal, must be using a highly effective contraception (including oral, transdermal, injectable, or implanted contraceptives, IUD, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 30 days prior to the first dose of OxabactTM and must agree to continue using such precautions during the clinical study.
19. Presence of a medical condition that the Principal Investigator considers likely to make the subject susceptible to adverse effect of study treatment or unable to follow study procedures. Note: Subjects from correctional facilities or asylums and subjects who are mentally handicapped are not to be included in the study.
20. Participation in any study of an investigational product, biologic, device, or other agent within 30 days prior to randomization or not willing to forego other forms of investigational treatment during this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in urinary oxalate levels (expressed as molar oxalate to creatinine ratio) from Baseline to Week 24 | 24 weeks

SECONDARY OUTCOMES:
Percentage change in urinary oxalate levels (expressed as molar oxalate to creatinine ratio) from Baseline to Week 8 | 8 weeks
Percentage change in urinary oxalate levels (expressed as molar oxalate to creatinine ratio) from Baseline to Week 24 in subsets of subjects defined by baseline urinary oxalate level, above and below median at screening | 24 weeks
Percentage change in urinary oxalate levels (expressed as molar oxalate to creatinine ratio) from Baseline to Week 24 in subsets of subjects defined by concomitant vitamin B6 therapy and no vitamin B6 therapy, in PH type I | 24 weeks
Percentage change in urinary oxalate levels (expressed as molar oxalate to creatinine ratio) from Baseline to Week 24 in subsets of subjects defined by eGFR of ≥90 mL/min/1.73m2 and < 90 mL/min/1.73m2 | 24 weeks
Percentage change in urinary oxalate levels (expressed as molar oxalate to creatinine ratio) from Baseline to Week 24 in subsets of subjects defined by PH Type I and PH Type II | 24 weeks
Percentage change in urinary oxalate levels (expressed as molar oxalate to creatinine ratio) from Baseline to Week 24 in subsets of subjects defined by age below 18 and age 18 or above | 24 weeks
Percentage of subjects who have ≥20% reduction from Baseline urinary oxalate at Week 24 | 24 weeks
Percentage change in plasma oxalate levels | 24 weeks
Frequency of Stone Events (i.e. nephrolithiasis or markers thereof) | 24 weeks
Correlation between percentage change in plasma oxalate levels and percentage change in urinary oxalate levels, from Baseline to Week 24 | 24 weeks
Adverse events (AEs), hematology, clinical chemistry, urinalysis. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Milliner, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- Mayo Clinic (Department of Pediatric Nephrology), Rochester, Minnesota, United States
- University Children's Hospital (Division of Pediatric Nephrology), Cologne, Germany
- Academy Medical Center, University of Amsterdam, Amsterdam, Netherlands